CLINICAL TRIAL: NCT03152162
Title: A Prospective Study to Evaluate the ConforMIS iTotal® (PS) Knee Replacement System
Status: Terminated | Type: Observational
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-003
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; patient-specific; knee replacement; TKA; knee arthroplasty; total knee replacement; posterior stabilized
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: iTotal PS KRS — Total knee arthroplasty for treatment of osteoarthritis
  Other Names: ConforMIS iTotal PS

SUMMARY:
This is a prospective clinical study designed to observe the long-term clinical outcomes of total knee arthroplasty using a patient-specific, posterior stabilized implant in patients with osteoarthritis.

DETAILED DESCRIPTION:
The study is prospective. Subjects will be implanted with an iTotal® PS Knee Replacement System. The study will include a minimum of 100 subjects across up to 10 sites. The patients enrolled in this study may represent the first cases of the iTotal PS KRS implanted at a particular site; data collected for the first 15 patients at each site will be analyzed separately from the rest of the enrolled population. This will provide visibility towards determining if there exists a learning curve in the implantation process of the iTotal PS KRS. The study sites will be located in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Clinical condition included in the approved Indications For Use for the iTotal® PS
* Osteoarthritis, as confirmed by the investigator's assessment of disease status at screening visit that warrants a TKR procedure. Disease status is assessed by Clinical and Radiographic assessment.
* Willingness to participate in the clinical study, to give informed consent, and to attend all follow-up visits
* > 18 years of age

Exclusion Criteria:

* Simultaneous bilateral procedure required
* BMI > 40
* Active malignancy (defined as a history of any invasive malignancy - except non- melanoma skin cancer), unless patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years
* Poorly controlled diabetes
* Neuromuscular conditions which prevent patient from participating in study activities
* Active local or systemic infection
* Immunocompromised
* Fibromyalgia or other general body pain related condition
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Loss of bone or musculature, osteonecrosis, neuromuscular or vascular compromise in the area of the joint to be operated on, to an extent that the procedure is unjustified
* Diagnosed with or receiving treatment for Osteoporosis
* Other physical disability affecting the hips, spine, or contralateral knee
* Severe instability due to advanced loss of osteochondral structure
* Prior arthroplasty of the affected knee, including High Tibial Osteotomy (HTO)
* Unwilling or unable to comply with study requirements
* Participation in another clinical study which would confound results
* Allergy to any of the implant materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarthritis of the knee
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Baseline from 1-Year in KSS | 2 Years
  Change in Knee Society Scores from the pre-operative visit to the 1-year post-operative visit. The Knee Society Score (KSS) includes an Objective Knee Score, Function Score, Satisfaction Score, and Expectation Score. The objective knee score, completed by the surgeon, includes a VAS score of pain walking on level ground and on stairs or inclines, as well as an assessment of alignment, ligament stability, and ROM, along with deductions for flexion contracture or extensor lag. Patients then record their satisfaction, functional activities, and expectations (Scuderi et al., 2012).

SECONDARY OUTCOMES:
Change from baseline in KSS at years 2, 5 and 10 post-implantation | Up to 10 years
  The Knee Society Score includes an Objective Knee Score, Function Score, Satisfaction Score, and Expectation Score. The Knee Society Score (KSS) includes an Objective Knee Score, Function Score, Satisfaction Score, and Expectation Score. The objective knee score, completed by the surgeon, includes a VAS score of pain walking on level ground and on stairs or inclines, as well as an assessment of alignment, ligament stability, and ROM, along with deductions for flexion contracture or extensor lag. Patients then record their satisfaction, functional activities, and expectations (Scuderi et al., 2012).
Change from baseline in KOOS at years 1, 2, 5 and 10 post-implantation | Up to 10 years
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a 42 question knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems.
Post-operative limb alignment if long leg x-rays available | 2 years
  Comparison of limb alignment between pre-operative and post-operative x-rays.
Length of hospital stay in hours | 1 year
  How long the patient is in the hospital from the time of admission to the time of discharge.
Blood loss during surgery | 1 year
  Estimated blood loss during surgery (mL)
Transfusion rate | 1 year
  Rate of patients who require blood transfusions during surgery

OTHER OUTCOMES:
Revision rates post-implantation | Collected from the date of implantation to the end of the study. Up to 10 years.
  Rate of patients that require a revision of the total knee replacement for any reason.
Length of procedure: Skin to Skin | 1 year
  The duration of the knee arthroplasty starting from the time the surgeon makes the first incision and ending when the surgeon sutures the initial incision.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quartulli, Study Director — Restor3D
Locations (4):
- United States (4):
  - UNC Orthopedics, Chapel Hill, North Carolina
  - Texas Institute for Hip & Knee Surgery, Austin, Texas
  - Mansfield Orthopaedics, Morrisville, Vermont
  - Scott Orthopedic, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Rougraff BT, Heck DA, Gibson AE. A comparison of tricompartmental and unicompartmental arthroplasty for the treatment of gonarthrosis. Clin Orthop Relat Res. 1991 Dec;(273):157-64. PMID 1959265
- [Background] Fitzpatrick C, FitzPatrick D, Lee J, Auger D. Statistical design of unicompartmental tibial implants and comparison with current devices. Knee. 2007 Mar;14(2):138-44. doi: 10.1016/j.knee.2006.11.005. Epub 2006 Dec 22. PMID 17188876
- [Background] Fitz W. Unicompartmental knee arthroplasty with use of novel patient-specific resurfacing implants and personalized jigs. J Bone Joint Surg Am. 2009 Feb;91 Suppl 1:69-76. doi: 10.2106/JBJS.H.01448. PMID 19182028
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035
- [Background] Scuderi GR, Bourne RB, Noble PC, Benjamin JB, Lonner JH, Scott WN. The new Knee Society Knee Scoring System. Clin Orthop Relat Res. 2012 Jan;470(1):3-19. doi: 10.1007/s11999-011-2135-0. No abstract available. PMID 22045067